CLINICAL TRIAL: NCT04285723
Title: Retrospective Chart Review Study of Patients With PIK3CA-Related Overgrowth Spectrum (PROS) Who Have Received Alpelisib as Part of a Compassionate Use Program (EPIK-P1)
Brief Title: Retrospective Chart Review Study of Patients With PIK3CA-Related Overgrowth Spectrum Who Have Received Alpelisib
Acronym: EPIK-P1
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CBYL719F12002
Record Dates: First submitted 2019-11-26; First posted 2020-02-26 (Actual); Results first posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2022-05

CONDITIONS: PIK3CA-Related Overgrowth Spectrum (PROS)
Keywords: alpelisib; PIK3CA; BYL719; PROS; Retrospective chart review study; EPIK-P1
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies | interventions — Alpelisib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- alpelisib: Patients treated with alpelisib
  Interventions: Other: alpelisib

INTERVENTIONS:
Other: alpelisib — Retrospective observational case-only study. There is no treatment allocation. Patients with severe or life-threatening PROS who have received alpelisib as part of a compassionate use program were invited to participate.

SUMMARY:
The study was a site-based retrospective non-interventional medical chart review of pediatric and adult male and female patients with PIK3CA-Related Overgrowth Spectrum (PROS) who initiated alpelisib at least 24 weeks before the cut-off date at a MAP site. The study cut-off date was 09-Mar-2020.

Patient-level data were abstracted from medical charts of all eligible patients at all participating sites. Study completion date refers to the last date data was extracted.

Information from patients treated with alpelisib was used to describe the efficacy and safety of alpelisib in PROS patients.

DETAILED DESCRIPTION:
The index date (baseline) is defined as the date of alpelisib initiation. The study period is the period from the index date up to the most recent data available at the time of the cut-off date.

The maximum follow-up was 187 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient (adult or pediatric) is ≥ 2 years of age
* Patient has a physician confirmed/documented diagnosis of PROS
* Patient has a documented evidence of a mutation in the PIK3CA gene
* Patient's condition was assessed by the treating physician as severe or life threatening and treatment was deemed necessary
* Patient has been treated with at least one dose of alpelisib, initiated on or before 23-Sep-2019 (i.e. at least 24 weeks before the cut-off date of the 09-Mar-2020)
* Patient has medical chart history available during enrollment in the Novartis MAP
* Patient (or parent/guardian in case of pediatric patient) consented to participate in the study (as required by local ethics regulations) Inclusion criteria for MAP enrollment (assessed at the time of alpelisib initiation)

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who participated in the compassionate use program and received alpelisib for the treatment of PIK3CA-related overgrowth spectrum (PROS).
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Boston Childrens Hospital, Boston, Massachusetts, United States
- Novartis Investigative Site, Parkville, Victoria, Australia
- France (3):
  - Novartis Investigative Site, Montpellier, Herault
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Paris
- Novartis Investigative Site, Dublin, Ireland
- Novartis Investigative Site, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fujino A, Kuniyeda K, Nozaki T, Ozeki M, Ohyama T, Sato I, Kamibeppu K, Tanaka A, Uemura N, Kanmuri K, Nakamura K, Kobayashi F, Suenobu S, Nomura T, Hayashi A, Nagao M, Kato A, Aramaki-Hattori N, Imagawa K, Ishikawa K, Ochi J, Horiuchi S, Nagabukuro H. The Prospective Natural History Study of Patients with Intractable Venous Malformation and Klippel-Trenaunay Syndrome to Guide Designing a Proof-of-Concept Clinical Trial for Novel Therapeutic Intervention. Lymphat Res Biol. 2024 Feb;22(1):27-36. doi: 10.1089/lrb.2023.0023. Epub 2023 Dec 19. PMID 38112724
- [Derived] Canaud G, Lopez Gutierrez JC, Irvine AD, Vabres P, Hansford JR, Ankrah N, Branle F, Papadimitriou A, Ridolfi A, O'Connell P, Turner S, Adams DM. Alpelisib for treatment of patients with PIK3CA-related overgrowth spectrum (PROS). Genet Med. 2023 Dec;25(12):100969. doi: 10.1016/j.gim.2023.100969. Epub 2023 Aug 24. PMID 37634128
- [Derived] Singh S, Bradford D, Li X, Mishra-Kalyani PS, Shen YL, Wang L, Zhao H, Xiong Y, Liu J, Charlab R, Kraft J, Khasar S, Miller CP, Rivera DR, Kluetz PG, Pazdur R, Beaver JA, Singh H, Donoghue M. FDA Approval Summary: Alpelisib for PIK3CA-Related Overgrowth Spectrum. Clin Cancer Res. 2024 Jan 5;30(1):23-28. doi: 10.1158/1078-0432.CCR-23-1270. PMID 37624421

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were from Australia (1), France (50), Ireland (1), Spain (3) and United States (2)
Groups:
- Pediatric Patients: Pediatric patients (< 18 years) treated with alpelisib
- Adult Patients: Adult patients (>= 18 years) treated with alpelisib
Period: Overall Study
Arm/Group | Pediatric Patients | Adult Patients
Started (Ful study population) | 39 | 18
Completed | 36 | 16
Not Completed | 3 | 2
Not completed — Subject decision | 1 | 2
Not completed — Physician Decision | 1 | 0
Not completed — No efficiency | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pediatric Patients | Adult Patients | Total
Number analyzed (Participants) | 39 | 18 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.9 (4.84) | 27.8 (8.34) | 15.5 (10.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 9 | 33
  Male | 15 | 9 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not reported | 32 | 18 | 50
  White | 7 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Responders and Non-responders at Week 24
Description: Response is defined by achieving at least 20% reduction from index date in the sum of measurable target lesion volume (1 to 3 lesions, via central review of imaging scans), provided that none of the individual target lesions have ≥ 20% increase from index date and in absence of progression of non-target lesions and without new lesions.
Time Frame: Index date and week 24 or 6 months (± 4 weeks)
Population: Efficacy population: It is a subset of the Full study population. It included patients with at least one target lesion and with an imaging scan performed on the index date (or up to 24 weeks prior to the index date) for at least one target lesion.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pediatric Patients | Adult Patients
Number analyzed (Participants) | 23 | 9
Percentage of participants
  Responders | 30.4 [13.2 to 52.9] | 55.6 [21.2 to 86.3]
  Non Responders | 69.6 [47.1 to 86.8] | 44.4 [13.7 to 78.8]

2. Secondary Outcome: Percent Change in the Sum of Measurable Target Lesion Volume
Description: Percent change in the sum of measurable target lesion (1 to 3 lesions) volume, as assessed by a central review of imaging scans, as measured by the change between the index date (or up to 24 weeks prior) and key time-points following the index date.
  The index date: (baseline) was defined as the date of alpelisib initiation End of study: patients were followed up to a maximum of 187 weeks.
Time Frame: Index date, week 4, 12 , 24, 52 and end of study (up to a maximum of week 187)
Population: Full study population: included all patients who satisfied the study inclusion criteria.
  At each time point, only patients with a value at both index date and that time point are included in the calculation of change
Measure: Mean (Standard Deviation); unit: % change in the sum of lesion vol.
Arm/Group | Pediatric Patients | Adult Patients
Number analyzed (Participants) | 22 | 9
% change in the sum of lesion vol.
  4 weeks: number analyzed (Participants) | 11 | 2
  4 weeks | -11.64 (12.869) | -11.78 (8.154)
  12 weeks: number analyzed (Participants) | 14 | 4
  12 weeks | -18.59 (16.837) | -19.77 (5.128)
  24 weeks | -11.20 (19.987) | -19.69 (15.375)
  52 weeks: number analyzed (Participants) | 16 | 4
  52 weeks | -13.91 (19.206) | -6.52 (2.614)
  End of study: number analyzed (Participants) | 4 | 3
  End of study | -36.47 (46.137) | -17.38 (11.679)

3. Secondary Outcome: Percent Change in the Sum of All Measurable Lesion Volume
Description: Percent change in the sum of all measurable (target and non-target) lesion volume, as assessed by a central review of imaging scans, as measured by the change between the index date (or up to 24 weeks prior) and key time-points following the index date.
  The index date (baseline) was defined as the date of alpelisib initiation. End of study: patients were followed up to a maximum of 187 weeks As no measurable non-target lesions were identified, the results for changes in the sum of all measurable (target and non-target) lesion volume were identical to the results presented for measurable target lesion.
Time Frame: Index date, week 4, 12 , 24, 52 and end of study (up to a maximum of week 187)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % change in the sum of lesion vol.
Arm/Group | Pediatric Patients | Adult Patients
Number analyzed (Participants) | 22 | 9
% change in the sum of lesion vol.
  4 weeks: number analyzed (Participants) | 11 | 2
  4 weeks | -11.64 (12.869) | -11.78 (8.154)
  12 weeks: number analyzed (Participants) | 14 | 4
  12 weeks | -18.59 (16.837) | -19.77 (5.128)
  24 weeks | -11.20 (19.987) | -19.69 (15.375)
  52 weeks: number analyzed (Participants) | 16 | 4
  52 weeks | -13.91 (19.206) | -6.52 (2.614)
  End of study: number analyzed (Participants) | 4 | 3
  End of study | -36.47 (46.137) | -17.38 (11.679)

4. Secondary Outcome: Percent Change in the Sum of All Measurable Non-target Lesion Volume
Description: Percent change in the sum of all measurable non-target lesion volume, as assessed by a central review of imaging scans, as measured by the change between the index date (or up to 24 weeks prior) and key time-points following the index date.
  The index date (baseline) was defined as the date of alpelisib initiation.
Time Frame: Index date, week 4, 12 , 24, 52 and end of study (up to a maximum of week 187)
Population: Full study population: included all patients who satisfied the study inclusion criteria. Only patients with non-target lesion are included in the analysis.
  Zero patients were included in this measure since no measurable non-target lesions were identified by independent central radiology review (ICRR) at the index date.
Arm/Group | Pediatric Patients | Adult Patients
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Mean Duration of Response (DoR)
Description: Duration of response is defined as the time from first documented response, to the date of the first documented disease progression or death due to any cause.
  Response is defined by achieving at least 20% reduction from index date in the sum of measurable target lesion volume (1 to 3 lesions, via central review of imaging scans), provided that none of the individual target lesions have ≥ 20% increase from index date and in absence of progression of non-target lesions and without new lesions.
  Disease progression is defined as an increase of any individual target lesions of ≥ 20% in volume from previous assessment, progression of non-target PIK3CA Related Overgrowth Spectrum (PROS) lesions or appearance of a new PROS lesion.
Time Frame: Up to 187 weeks
Population: Efficacy population: It is a subset of the Full study population. This analysis only applied to responders with documented disease progression or death due to any cause.
Arm/Group | Pediatric Patients | Adult Patients
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Reasons for Discontinuation of Concomitant PROS-related Non-drug Treatments
Description: Number of participants with concomitant PIK3CA Related Overgrowth Spectrum (PROS)-related non-drug treatments and other medical interventions by reason for discontinuation.
  A patient may have multiple information, but was counted only once in type of other supportive non-drug treatment if more than one type in this category has been reported.
Time Frame: Up to 187 weeks
Population: Full study population: included all patients who satisfied the study inclusion criteria. Only patients who were under concomitant PROS-related non-drug treatments were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Patients | Adult Patients
Number analyzed (Participants) | 31 | 17
Participants
  Recovery | 12 | 2
  Completed the planned course of treatment | 4 | 7
  Unknown | 2 | 1
  Lack of efficacy | 1 | 1
  Other | 2 | 0
  Adverse event | 0 | 1
  Progressive disease | 0 | 1
  Subject decision | 0 | 1

7. Secondary Outcome: Participants With Concomitant PROS-related Medications Over Time
Description: Number of participants with at least one concomitant utilization of PIK3CA Related Overgrowth Spectrum (PROS)-related medication.
  End of study: patients were followed up to a maximum of 187 weeks. Results are provided for the full study population as planned and documented in the protocol and SAP, and not by age group.
Time Frame: Index date, week 24 and end of study
Population: Full study population: included all patients who satisfied the study inclusion criteria.
Measure: Count of Participants; unit: Participants
Groups:
- All Patients: Pediatric and adult patients treated with alpelisib
Arm/Group | All Patients
Number analyzed (Participants) | 57
Participants
  Index date | 34
  24 weeks: number analyzed (Participants) | 56
  24 weeks | 30
  End of study | 25

8. Secondary Outcome: Number of PROS-related Completed Surgeries During the Study Period
Description: Number of surgeries by reason of surgery. A patient may have multiple anatomical sites of surgery and types of surgery on the same day.
Time Frame: Up to 187 weeks
Population: Full study population: included all patients who satisfied the study inclusion criteria.
Measure: Number; unit: Surgeries
Arm/Group | Pediatric Patients | Adult Patients
Number analyzed (Participants) | 39 | 18
Surgeries
  Other | 4 | 2
  Disease improvement | 2 | 1
  Disease progression (not radiologically confirmed) | 3 | 0

9. Secondary Outcome: Number of Patients With Improvement in Most Frequent PROS-related Signs and Symptoms
Description: Improvement in PIK3CA Related Overgrowth Spectrum (PROS) signs and symptoms was defined based on Common Toxicity Criteria (CTC) grade reduction or resolution of the event from index date.
  CTC is a set of criteria for the standardized classification of adverse effects of drugs used in cancer therapy. The Common Terminology Criteria for Adverse Events (CTCAE) system is a product of the US National Cancer Institute (NCI). For this study, version 4.03 was used
Time Frame: Index date and week 24 or 6 months (± 4 weeks)
Population: Full study population: included all patients who satisfied the study inclusion criteria. For the assessment of improvement for the individual items, only patients with the symptom at the index date were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Patients | Adult Patients
Number analyzed (Participants) | 39 | 18
Participants
  Fatigue improved by week 24: number analyzed (Participants) | 28 | 14
  Fatigue improved by week 24 | 22 | 10
  Vascular malformation improved by week 24: number analyzed (Participants) | 25 | 13
  Vascular malformation improved by week 24 | 20 | 10
  Disseminated intravascular coagulation improved by week 24: number analyzed (Participants) | 19 | 10
  Disseminated intravascular coagulation improved by week 24 | 11 | 5
  Limb asymmetry improved by week 24: number analyzed (Participants) | 17 | 12
  Limb asymmetry improved by week 24 | 11 | 9
  Pain improved by week 24: number analyzed (Participants) | 12 | 10
  Pain improved by week 24 | 11 | 9

10. Secondary Outcome: Change in Performance Status Score
Description: Participants with a change in performance status score (ECOG, Karnofsky, Lansky) between the index date and week 24. Patients completed one questionnaire (ECOG, Karnofsky or Lansky) based on physicians choice.
  The Eastern Cooperative Oncology Group (ECOG) score runs from 0 to 5, with 0 denoting perfect health and 5 death. The Karnofsky Performance Score (KPS) and Lansky score run from 0 to 100, where 0 is death and 100 is perfect health.
  For the ECOG scale, "improvement" is defined as a decrease by at least 1 point and and "worsening" is defined as an increase by at least 1 point. For the Karnofsky and Lansky scale, "improvement" is defined as an increase by at least 20 points and worsening is defined as a decrease by at least 20 points.
  If neither of the criteria for improvement or worsening is met, then it is considered stable.
Time Frame: Index date and week 24 or 6 months (± 4 weeks)
Population: Full study population: included all patients who satisfied the study inclusion criteria.
  Only patients with performance status (ECOG, Karnofsky, Lansky) assessed at the index date were included in the calculation of change
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Patients | Adult Patients
Number analyzed (Participants) | 33 | 14
Participants
  Stable | 9 | 1
  Improved | 8 | 6
  Worsened | 0 | 0
  Not reported | 16 | 7

11. Secondary Outcome: Functional Status - Mobility Assessment
Description: Change in functional status: Mobility severity assessment measured up to the judgment of the investigator.
  A patient may have multiple information
Time Frame: Up to 187 weeks
Population: Full study population: included all patients who satisfied the study inclusion criteria.
  Only patients with at least one mobility assessment were included in the severity assessment.
Measure: Count of Units; unit: Affected regions
Units Other Than Participants: Affected regions
Arm/Group | Pediatric Patients | Adult Patients
Number analyzed (Participants) | 1 | 2
Number analyzed (Affected regions) | 1 | 6
Affected regions
  No impairment | 0 | 1
  Mild impairment | 0 | 1
  Moderate impairment | 1 | 2
  Severe impairment | 0 | 1
  Missing | 0 | 1

12. Secondary Outcome: Change From Index Date in Functional Status - School Status During the Study Period
Description: Change in functional status: School status during the study period (no attendance, part-time or full time).
  Improvement is defined as a shift from reporting of "No attendance" to "Part-time" as well as , "Part-time" or "No attendance" to "Full-time"; Worsening is defined as a shift from reporting of "Part-time" to "No attendance", as well as from "Full-time" to "Part-time" or "No attendance".
  If neither of the criteria for improvement or worsening is met, then it is considered stable.
Time Frame: Index date, week 24 and end of study (up to 187 weeks)
Population: Full study population: included all patients who satisfied the study inclusion criteria.
  Only patients reporting school status at index date were included in the calculation of change
Measure: Count of Participants; unit: Participants
Groups:
- Pediatric Patients: Pediatric patients (< 18 years) treated with alpelisib reporting school status
- Adult Patients: Adult patients (>= 18 years) treated with alpelisib reporting school status
Arm/Group | Pediatric Patients | Adult Patients
Number analyzed (Participants) | 29 | 4
Participants
  Change 24 weeks: Improvement | 1 | 0
  Change 24 weeks: Stable | 28 | 4
  Change 24 weeks: missing | 0 | 0
  Change 24 weeks: Worsening | 0 | 0
  End of study: Improvement | 2 | 2
  End of study: Stable | 27 | 2
  End of study: missing | 0 | 0
  End of study: Worsening | 0 | 0

13. Secondary Outcome: Change From Index Date in Functional Status - Work Status
Description: Change in functional status: Work status assessment during the study period (no attendance, part-time, full-time or unemployed).
  Improvement is defined as a shift from reporting of "No attendance" to "Part-time" or "Full time", from "Part-time" to "Full-time", as well as from "Unemployed" to "Part-time" or "Full-time" work.
  Worsening is defined as a shift from reporting of "Part-time" to "No attendance", "Full-time" to "Part-time" or "No attendance" as well as "Part-time" or "Full-time" to "Unemployed" status.
  Change in score is only applicable if both index date and post-index date information are available.
  If a patient has more than 1 score reported within the same time window, the worst is considered.
  If neither of the criteria for improvement or worsening is met, then it is considered stable.
Time Frame: Index date, week 24 and end of study
Population: Full study population: included all patients who satisfied the study inclusion criteria.
  Only adult patients reporting work status at index date were included in the calculation of change.
Measure: Count of Participants; unit: Participants
Groups:
- Adult Patients: Adult patients (>= 18 years) treated with alpelisib reporting work status
Arm/Group | Adult Patients
Number analyzed (Participants) | 8
Participants
  Change 24 weeks: Improvement | 0
  Change 24 weeks: Worsening | 1
  Change 24 weeks: Stable | 6
  Change 24 weeks: Missing | 1
  Change end of study: Improvement | 5
  Change end of study: Worsening | 0
  Change end of study: Stable | 2
  Change end of study: Missing | 1

14. Secondary Outcome: Health Resource Utilization (HRU) - Number of Hospitalizations Per Patient
Description: Hospitalizations starting on or after the start of study treatment (index date) or starting prior to and continuing after the start of study treatment are summarized.
Time Frame: Up to 187 weeks
Population: Full study population: included all patients who satisfied the study inclusion criteria.
Measure: Mean (Standard Deviation); unit: Number of hospitalizations
Arm/Group | Pediatric Patients | Adult Patients
Number analyzed (Participants) | 39 | 18
Number of hospitalizations
  Number of times a patient has been hospitalized | 1.8 (1.03) | 1.7 (0.82)
  Number of times a patient has been hospitalized due to PROS | 1.1 (0.35) | 1.0 (0.00)

15. Secondary Outcome: Number of Patients With Grade 3/4 on Laboratory Assessments: Hematology
Description: Worst post-index date hematology abnormalities based on Common Toxicity Criteria (CTC) grades during the study period.
  Grade refers to the severity of the AE: Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living. Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living. Grade 4 Life-threatening consequences; urgent intervention indicated.
  Patients are counted only for the worst grade observed post-index date values. Laboratory assessments performed more than 30 days after last study treatment administration date are not summarized.
Time Frame: Up to 187 weeks
Population: Full study population: included all patients who satisfied the study inclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Patients | Adult Patients
Number analyzed (Participants) | 39 | 18
Participants
  Activated partial thromboplastin time, increase - Grade 3/4 | 0 | 0
  Fibrinogen, decrease - Grade 3/4 | 0 | 0
  Hemoglobin, decrease - Grade 3/4 | 2 | 1
  Leukocytes, increase - Grade 3/4 | 1 | 0
  Leukocytes, decrease - Grade 3/4 | 0 | 0
  Lymphocytes, increase - Grade 3/4 | 0 | 0
  Lymphocytes, decrease - Grade 3/4 | 0 | 1
  Neutrophils, decrease - Grade 3/4 | 0 | 1
  Platelets, decrease - Grade 3/4 | 0 | 1

16. Secondary Outcome: Number of Patients With Grade 3/4 on Clinical Assessments - Clinical Chemistry
Description: Worst post-index date biochemistry abnormalities based on Common Toxicity Criteria (CTC) grades.
  Grade refers to the severity of the AE: Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living. Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living. Grade 4 Life-threatening consequences; urgent intervention indicated.
  Patients are counted only for the worst grade observed post-index date values. Laboratory assessments performed more than 30 days after last study treatment administration date are not summarized.
Time Frame: 187 weeks
Population: Full study population: included all patients who satisfied the study inclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Patients | Adult Patients
Number analyzed (Participants) | 39 | 18
Participants
  Alanine Aminotransferase Increase - Grade 3/4 | 0 | 0
  Albumin Decrease - Grade 3/4 | 0 | 0
  Alkaline Phosphatase Increase - Grade 3/4 | 0 | 0
  Aspartate Aminotransferase Increase - Grade 3/4 | 0 | 0
  Bilirubin Increase - Grade 3/4 | 0 | 2
  Calcium Corrected Increase - Grade 3/4 | 0 | 0
  Calcium Corrected Decrease - Grade 3/4 | 0 | 0
  Cholesterol Increase - Grade 3/4 | 0 | 0
  Creatine Kinase Increase - Grade 3/4 | 0 | 0
  Creatinine Increase - Grade 3/4 | 0 | 0
  Gamma Glutamyl Transferase Increase - Grade 3/4 | 0 | 0
  Glucose Increase - Grade 3/4 | 0 | 1
  Magnesium Increase - Grade 3/4 | 1 | 0
  Magnesium Decrease - Grade 3/4 | 0 | 1
  Phosphate Decrease - Grade 3/4 | 0 | 2
  Potassium Increase - Grade 3/4 | 0 | 0
  Potassium Decrease - Grade 3/4 | 0 | 0
  Sodium Increase - Grade 3/4 | 0 | 0
  Sodium Decrease - Grade 3/4 | 0 | 1
  Triglycerides Increase - Grade 3/4 | 0 | 0
  Urate Increase - Grade 3/4 | 1 | 1

17. Secondary Outcome: Notable Vital Sign Values During the Study Period - Pediatric Patients
Description: Low/High: Indicating abnormal value/change from index date.
  High systolic blood pressure: ≥95th percentile of the age and height group Low Systolic blood pressure: ≤5th percentile of the age and height group. High diastolic blood pressure: ≥95th percentile of the age and height group Low diastolic blood pressure: ≤5th percentile of the age and height group. High pulse rate (bpm): 2-3 years: >128; 3-4 years: >123; 4-6 years: >117; 6-8 years: >111; 8-12years: >103; 12-15 years: >96; ≥15 years: >92 Low pulse rate (bpm): 2-3 years: <92; 3-4 years: <86; 4-6 years: <81; 6-8 years: <74; 8-12 years: <67; 12-15 years: <62; ≥15 years: <58.
  High weight: increase from baseline of ≥2 Body mass index (BMI) for age percentile categories Low weight: decrease from baseline of ≥2 BMI-for-age percentile categories
Time Frame: End of study (up to week 187)
Population: Full study population: included all patients who satisfied the study inclusion criteria. Only pediatric patients were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Patients
Number analyzed (Participants) | 35
Participants
  High Systolic blood pressure | 17
  Low Systolic blood pressure | 3
  High Diastolic blood pressure | 12
  Low Diastolic blood pressure | 2
  High Pulse rate: number analyzed (Participants) | 34
  High Pulse rate | 15
  Low Pulse rate: number analyzed (Participants) | 34
  Low Pulse rate | 10
  High Weight: number analyzed (Participants) | 29
  High Weight | 0
  Low Weight: number analyzed (Participants) | 29
  Low Weight | 1

18. Secondary Outcome: Notable Vital Sign Values During the Study Period - Adult Patients
Description: Low/High: Indicating abnormal value/change from index date.
  High systolic blood pressure: ≥180 mmHg and increase ≥20 mmHg Low systolic blood pressure: ≤90 mmHg and decrease ≥20 mmHg. High diastolic blood pressure: ≥105 mmHg and increase ≥15 mmHg Low diastolic blood pressure: ≤50 mmHg and decrease ≥15 mmHg. High pulse rate: ≥120 bpm and increase ≥15 bpm Low pulse rate: ≤ 50 bpm and decrease ≥15 bpm. High weight: Increase ≥10% Low weight: Decrease ≥10%
Time Frame: End of study (up to week 187)
Population: Full study population: included all patients who satisfied the study inclusion criteria. Only adult patients were included in this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Patients | Adult Patients
Number analyzed (Participants) | 35 | 17
Participants
  High Systolic blood pressure | 17 | 0
  Low Systolic blood pressure | 3 | 0
  High Diastolic blood pressure | 12 | 2
  Low Diastolic blood pressure | 2 | 0
  High Pulse rate: number analyzed (Participants) | 34 | 17
  High Pulse rate | 15 | 1
  Low Pulse rate: number analyzed (Participants) | 34 | 17
  Low Pulse rate | 10 | 0
  High Weight: number analyzed (Participants) | 29 | 15
  High Weight | 0 | 0
  Low Weight: number analyzed (Participants) | 29 | 15
  Low Weight | 1 | 6

19. Secondary Outcome: Number of Participants With Notable ECG Values.
Description: Notable Electrocardiogram (ECG) values during the study period
Time Frame: Up to week 187
Population: Full study population: included all patients who satisfied the study inclusion criteria. Only patients with ECG data are included in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Pediatric Patients: Pediatric patients (< 18 years) treated with alpelisib reporting ECG values
- Adult Patients: Adult patients (>= 18 years) treated with alpelisib reporting ECG values
Arm/Group | Pediatric Patients | Adult Patients
Number analyzed (Participants) | 3 | 3
Participants
  QTcF New >450 to <=480 ms: number analyzed (Participants) | 3 | 2
  QTcF New >450 to <=480 ms | 1 | 1
  QT Increase >30 to <=60 ms: number analyzed (Participants) | 3 | 1
  QT Increase >30 to <=60 ms | 1 | 0
  QT New >480 to <=500 ms | 0 | 1

20. Secondary Outcome: Growth and Development in Pediatric Population
Description: Assessed in patients who were aged <18 years at the time of alpelisib initiation.
  SDS (standard deviation scores) for height and BMI are obtained from the WHO Growth Charts, and SDS for height and weight velocity are obtained from Baumgartner et al. (1986). Height or weight velocity is a variable derived from the measurement of height or weight at different times and represents the increase in height or weight during a fixed period.
  SD- scores are used to describe how far a measurement is from the median (average).
  Weight-for-age reference data are not available beyond age 10.
Time Frame: Week 24 or 6 months (± 4 weeks)
Population: Full study population: included all pediatric patients who satisfied the study inclusion criteria. Only patients with SD-score available are included.
Measure: Mean (Standard Deviation); unit: SD-score
Arm/Group | Pediatric Patients
Number analyzed (Participants) | 29
SD-score
  Height SDS | -0.1 (1.23)
  Height velocity SDS: number analyzed (Participants) | 26
  Height velocity SDS | 0.1 (5.01)
  BMI SDS: number analyzed (Participants) | 26
  BMI SDS | 0.8 (1.21)
  Weight velocity SDS: number analyzed (Participants) | 16
  Weight velocity SDS | -0.2 (2.86)

21. Secondary Outcome: Overview of Number of Patients With Adverse Events (AEs)
Description: A patient with multiple severity grades for an AE is only counted under the maximum grade.
  All grades includes any AEs with missing grade. Grade refers to the severity of the AE: Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living. Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living. Grade 4 Life-threatening consequences; urgent intervention indicated.
Time Frame: Up to 187 weeks
Population: Full study population: included all patients who satisfied the study inclusion criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Patients | Adult Patients
Number analyzed (Participants) | 39 | 18
Participants
  Adverse events - All grades | 31 | 16
  Adverse events - Grade ≥ 3 | 4 | 9
  SAEs - All grades | 10 | 11
  SAEs - Grade ≥ 3 | 3 | 9
  AEs leading to dose reduction - All grades | 0 | 3
  AEs leading to dose reduction - Grade ≥ 3 | 0 | 0
  AEs leading to dose interruption - All grades | 2 | 3
  AEs leading to dose interruption - Grade ≥ 3 | 0 | 2
  AEs leading to treatment discontinuation | 0 | 0
  SAEs treatment-related - All grades | 0 | 3
  SAEs treatment-related - Grade ≥ 3 | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment or cut-off date whichever occurs first, up to maximum duration of 187 weeks
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment or cut-off date whichever occurs first
Arm/Group | Pediatric Patients | Adult Patients
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/18
Serious Adverse Events (participants affected / at risk) | 10/39 | 11/18
Other Adverse Events (participants affected / at risk) | 23/39 | 16/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pediatric Patients (N=39) | Adult Patients (N=18)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Vascular malformation (Congenital, familial and genetic disorders) | 2 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Volvulus (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Gait disturbance (General disorders) | 2 | 0
Impaired healing (General disorders) | 0 | 1
Inflammation (General disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 0
Otitis media acute (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 | 0
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypotonia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pediatric Patients (N=39) | Adult Patients (N=18)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 | 2
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1
Vascular malformation (Congenital, familial and genetic disorders) | 2 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 3 | 3
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 4
Haemorrhoids (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 0
Toothache (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
Inflammation (General disorders) | 3 | 1
Abscess soft tissue (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Prostatitis Escherichia coli (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 2 | 0
Weight decreased (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Folate deficiency (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 0 | 3
Memory impairment (Nervous system disorders) | 0 | 2
Sciatica (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1
Libido decreased (Psychiatric disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Haematospermia (Reproductive system and breast disorders) | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Vaginal ulceration (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 3
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 3
Eczema (Skin and subcutaneous tissue disorders) | 1 | 3
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 2
Haematoma (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/23/NCT04285723/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/23/NCT04285723/SAP_001.pdf